CLINICAL TRIAL: NCT05265130
Title: Evaluation of Efficacy of YiQiFuMai Injection as an Adjunctive Treatment for Sepsis: a Single Center Randomized Controlled Pilot Study
Brief Title: The Efficacy of YiQiFuMai Injection as an Adjunctive Treatment for Sepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Anlu Wang, MD, Prof., Xiyuan Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI2021A02908
Record Dates: First submitted 2021-12-26; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — yi-qi-fu-mai; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YQFM group (Experimental): YQFM 5.2g in 0.9% Normal Saline 250ml IV, about 40 drops per min, once a day.
  Interventions: Drug: YiQiFuMai
- Placebo group (Placebo Comparator): 0.9% Normal Saline 250ml IV, about 40 drops per min.
  Interventions: Drug: 0.9% Normal Saline 250ml

INTERVENTIONS:
Drug: YiQiFuMai — YQFM is a redeveloped preparation based on the traditional Chinese medicine formula Sheng-Mai-San, which is widely used in clinical practice in China, mainly for the microcirculatory disturbance-related diseases.
  Arms: YQFM group
Drug: 0.9% Normal Saline 250ml — 0.9% Normal Saline 250ml IV, about 40 drops per min.
  Arms: Placebo group

SUMMARY:
This is a prospective single center pilot randomized controlled study to assess the efficacy and safety of YiQiFuMai injection (YQFM), a widely used Chinese medicine, as an adjunctive treatment for sepsis.

DETAILED DESCRIPTION:
Sepsis is a major clinical challenge with high mortality and morbidity worldwide. Sepsis is characterized by the dysregulated host response to an infection followed by organ dysfunction. Early sepsis mortality has diminished with advances in intensive care management and goal-directed interventions, only to surge after "recovery" from acute events, which prompts a search for sepsis-induced alterations in immune function. When suffered from sepsis, patients may have evidence of hyper-inflammation and immunosuppression. There are no high-quality evidence examining the effect of intravenous (IV) immunoglobulins or other immune modulators on the outcomes of patients with sepsis or septic shock. YiQiFuMai Injection (YQFM) is a redeveloped preparation based on the traditional Chinese medicine formula Sheng-Mai-San, which is widely used in clinical practice in China, mainly for the microcirculatory disturbance-related diseases. YQFM is proved to be effective for treating sepsis (unpublished data). And several researches reveal that YQFM attenuates acute respiratory distress syndrome and lipopolysaccharide-induced microvascular disturbance in vitro.

The purpose of this study is to explore the adjunctive treatment effect of YQFM to prognosis, immune dysfunction and organ dysfunction of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis defined by Sepsis-3 definition
* Adult patients between the ages of 18 and 90.
* Informed consent is provided by patients or obtained by family member if patient is incapacitated.

Exclusion Criteria:

* Known severe allergic reaction to drugs including but not limited to YQFM.
* Pregnant patients or those who may be pregnant
* Patients with severe intracranial diseases (intracranial artery stenosis, intracranial infection, cerebral hemorrhage, cerebral infarction, brain trauma, subjects after intracranial surgery)
* Patients with extremely severe brain injury, after cardiopulmonary resuscitation, advanced malignant tumor, combined with serious primary diseases such as liver, lung, kidney and hematopoietic system, and poor prognosis;
* Autoimmune diseases, immune deficiency diseases, continuous use of immunosuppressants within the last 6 months, or organ transplants;
* Major surgery or trauma within the last 2 weeks;
* Participated in other clinical trials or took similar drugs within 1 month;
* The investigator considered that the subjects had poor compliance or other clinical, social, or family factors that were inappropriate for inclusion in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
All-cause Mortality [28 days after randomization] | In 28 days after randomization
  Death from all causes at 28-days
Mortality in ICU and several time points | In 14 days after randomization
  Death from all causes at ICU discharge, 7 days, and 14 days after randomization
The secondary infection rate in 28 days. | In 28 days after randomization
Length of stay in ICU | up to 28 days after randomization
Absolute lymphocyte count in the routine blood test (*10^9g/L) | Change from baseline at 14 days after randomization
Concentration of T cells and B cells | Change from baseline at 14 days after randomization
  CD3+CD4-CD8-, CD3+CD4+CD8-, CD3+CD4-CD8+, CD3+CD4+CD8+, CD3+CD19-, CD3-CD19+, CD3+(CD16+CD56)+, CD3-(CD16+CD56)+ ,CD4+CD25+,CD4+CD25+CD127- (cells/uL)
Concentration of inflammatory cytokines | Change from baseline at 14 days after randomization
  interleukin (IL) 1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-17, interferon (IFN) α, IFN-γ, and Tumor nuclear factor (TNF)-α. (pg/mL);
Concentration of Procalcitonin | Change from baseline at 14 days after randomization
Length of stay in hospital | up to 28 days after randomization

SECONDARY OUTCOMES:
Duration of mechanical ventilation (MV) in ICU | up to 28 days after randomization
Duration of continual renal replacement therapy (CRRT) in ICU | up to 28 days after randomization
Duration of vasopressor drugs in ICU | up to 28 days after randomization
Duration of fluid resuscitation in ICU | up to 28 days after randomization
Total amount of fluid resuscitation (mL) in ICU | up to 28 days after randomization
SOFA score | Change from baseline at 14 days after randomization
  Total Sequential Organ Failure Assessment (SOFA) score (0-24), higher values represent a worse outcome
APACHEII | change from baseline at 7 days after randomization
  Acute Physiology and Chronic Health Evaluation (include Acute physiology score, APS and age and Chronic physiology score, totally 0-71 Points)
Self-Rating Anxiety Scale (SAS) score | change from baseline at 28 days after randomization
  Score range from 0 to 80, higher values represent a worse outcome
Self-Rating Depression Scale (SDS) score | change from Day 7 at 28 days after randomization
  Score range from 0 to 80, higher values represent a worse outcome
Barthel score | change from baseline at 28 days after randomization
  Score range from 0 to 100, higher values represent a better outcome
The mean artery pressure (MBP) | change from baseline at 7 days after randomization
The worst heart rate | change from baseline at 7 days after randomization
Concentration of serum lactate | change from baseline at 14 days after randomization
The rate of lactate clearance | change from baseline at 14 days after randomization
  (baseline lactate-lactate)/baseline lactate
The volume of urine output | change from baseline at 14 days after randomization
Concentration of IgM, IgG, IgE (g/L) (blood) | change from baseline at 14 days after randomization
Concentration of complement in serum (C3 and C4) (g/L) | change from baseline at 14 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zhixu Yang, Prof., Principal Investigator — Xiyuan Hospital

IPD SHARING:
Plan to Share IPD: No